CLINICAL TRIAL: NCT04325009
Title: A Open-Label, Randomized, 2-sequence, 4-period, Fasting Condition, Singledose, Per Oral, Cross-over Study to Evaluate the Bioequivalence Between "Dong-A Atorvastatin 80mg Tab" and "Lipitor 80mg Tab" in Healthy Volunteers
Brief Title: Bioequivalence Study Between "Dong-A Atorvastatin Tab" and "Lipitor Tab"
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DDS19-066BE
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Crossover Assignment single-dose, 2-sequence, 4-period Bioequivalence Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTRT (Experimental): R: "Lipitor 80mg Tab" T: "Dong-A Atorvastatin 80mg Tab"
  Interventions: Drug: Lipitor 80mg Tab → Dong-A Atorvastatin 80mg Tab
- TRTR (Experimental): R: "Lipitor 80mg Tab" T: "Dong-A Atorvastatin 80mg Tab"
  Interventions: Drug: Dong-A Atorvastatin 80mg Tab → Lipitor 80mg Tab

INTERVENTIONS:
Drug: Lipitor 80mg Tab → Dong-A Atorvastatin 80mg Tab — 1. st period: single oral administration of 1 tablet of "Lipitor 80mg Tab" washout period: 7days
  2. nd period: single oral administration of 1 tablet of "Dong-A Atorvastatin 80mg Tab" washout period: 7days
  3. rd period: single oral administration of 1 tablet of "Lipitor 80mg Tab" washout period: 7days
  4. th period: single oral administration of 1 tablet of "Dong-A Atorvastatin 80mg Tab"
  Arms: RTRT
Drug: Dong-A Atorvastatin 80mg Tab → Lipitor 80mg Tab — 1. st period: single oral administration of 1 tablet of "Dong-A Atorvastatin 80mg Tab" washout period: 7days
  2. nd period: single oral administration of 1 tablet of "Lipitor 80mg Tab" washout period: 7days
  3. rd period: single oral administration of 1 tablet of "Dong-A Atorvastatin 80mg Tab" washout period: 7days
  4. th period: single oral administration of 1 tablet of "Lipitor 80mg Tab"
  Arms: TRTR

SUMMARY:
An Open-Label, Randomized, 2-sequence, 4-period, Fasting Condition, Single-dose, Per Oral, Cross-over Study to Evaluate the Bioequivalence between "Dong-A Atorvastatin 80mg Tab" and "Lipitor 80mg Tab" in Healthy Volunteers

DETAILED DESCRIPTION:
1. Study design: An open-Label, randomized, 2-sequence, 4-period, fasting condition, single-dose, per oral, cross-over study
2. Administration method:

   The subject should maintain a minimum of 10 hours of empty stomach before administration, and give an oral dose of 1 tablets (Dong-A Atorvastatin 80mg or Lipitor 80mg) with 150 mL of water at around 8 a.m. on the day of the test. The subject should not chew or break the drug, but should swallow in whole with water. The difference in administration time between the test subjects is about one minute apart, considering the blood collection time.
3. Wash out period: at least 7 days
4. Blood collection time: Before the administration, 0.17, 0.33, 0.5, 0.75, 1, 1.33, 1.67, 2, 3, 4, 6, 8, 12, 24, 36 hr after the administration (total 16 times)
5. Analysis: Measurement of the concentration of an unchangeable substance of Atorvastatin in plasma

ELIGIBILITY:
Inclusion Criteria:

1. A person who aged 19 or older at the time of screening
2. BMI of 18 to 30 (BMI calculation: kg/m2)

   * Males weighing 50kg or more
   * Females weighing 45kg or more
3. No congenital or chronic diseases or pathological symptoms
4. A person who is judged to be suitable for the study by the investigator based on the clinical laboratory examination
5. A person who has fully understood the contents of the consent form for the study and signed the consent form voluntarily and recorded the date of signature
6. A person who agreed to use contraception from the first administration of IP to a week after the last administration of IP

Exclusion Criteria:

1. A person who has taken a drug that significantly induces (e.g., barbital) or inhibits the drug metabolic enzyme within 30 days prior to the first administration of IP
2. A person who has participated in other clinical trials within six months prior to the first administration of the IP
3. A person who has had whole blood transfusion within 2 months or the apheresis within 2 weeks before the first administration of IP
4. A person who has medical history of gastric resection that can affect the drug absorption
5. A person with a history of regular alcohol intake within a month prior to the first administration of the IP:

   * Male: More than 21 cups/week
   * Female: More than 14 cups/week (1 cup: 50 ml of soju, 250 ml of beer, 30ml of spirits)
6. A person who is hypersensitive to any of the IP components, taking glecaprevir, pibrentasvir, has active hepatic disease, Blood AST (GOT) or ALT (GPT) levels exceed the upper reference range limit by 3 times, muscle disease, or any genetic symtoms such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
7. A person who has medical history of mental disease
8. A person who is judged not to be suitable for the study by the investigator
9. Lactating or possibly pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Area Under the plasma Concetration versus time curve(AUCt) of Atorvastatin | Before administration ~ 36hrs
  Area Under the plasma Concetration versus time curve(AUCt) of Atorvastatin
Peak Plasma Concentration(Cmax) of Atorvastatin | Before administration ~ 36hrs
  Peak Plasma Concentration(Cmax) of Atorvastatin

CONTACTS AND LOCATIONS:
Overall Officials: SeungHyun Kang, Ph.D, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea